CLINICAL TRIAL: NCT05099757
Title: The Study on the Immunogenicity and Persistence of Booster Dose With Hepatitis B Vaccine in College Students
Brief Title: The Immunogenicity and Persistence of Booster Dose With Hepatitis B Vaccine in College Students
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Suping Wang, Professor, Shanxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DXSHB20211012
Record Dates: First submitted 2021-10-13; First posted 2021-10-29 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis B Vaccine
Keywords: Hepatitis B Vaccine; Immunogenicity; Booster Dose; Long-term Immune Response; College Students
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20 µg at month 0, months 0, 1 or 0, 1, and 6 (Experimental): 20 µg recombinant hepatitis B vaccine with one, two or three injections at month 0, months 0, 1 or 0, 1, and 6
  Interventions: Biological: 20 µg dose hepatitis B vaccine

INTERVENTIONS:
Biological: 20 µg dose hepatitis B vaccine — one-dose, two-dose or three-dose, 20 µg per dose

SUMMARY:
The anti-HBs produced after hepatitis B vaccination will decrease over time. College students are vaccinated with hepatitis B vaccine at birth, and their antibodies may have decreased significantly. In addition, college students are sexually active population, which has a high risk of HBV infection. It is necessary to study the anti-HBs level of college students, and analyze the strengthening immunization for this special group.

This study will analyze the immunogenicity, immune persistence, and safety of booster dose of intramuscular 20 µg recombinant hepatitis B vaccines. Different booster vaccination including one-dose (0 month), two-dose (0, 1 months), or three-dose (0, 1, and 6 months) was given according to the antibody production level after booster vaccination among college students.

DETAILED DESCRIPTION:
Participants are given booster dose of one-dose (0 month), two-dose (0, 1 months), or three-dose (0, 1, and 6 months) 20 µg recombinant hepatitis B vaccine according to the antibody production level. HBsAg and anti-HBs will be tested during the study period. Adverse reactions will be recorded after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged of 18 years or above
* Serologically negative for hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (anti-HBs) at enrollment
* Sign informed consent, willing to participate in this study

Exclusion Criteria:

* Being pregnant
* Intolerance or allergy to any component of the vaccine
* Participants with severe acute or chronic diseases (such as liver disease, blood disease, cancer), acute onset of chronic diseases and fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2022-11-25 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Anti-HBs Seroconversion Rate at Months 1 | Months 1
  Anti-HBs Seroconversion Rate at Months 1
Anti-HBs Seroconversion Rate at Months 3 | Months 3
  Anti-HBs Seroconversion Rate at Months 3
Anti-HBs Seroconversion Rate at Months 7 | Months 7
  Anti-HBs Seroconversion Rate at Months 7
Anti-HBs Seroconversion Rate at Months 12 | Months 12
  Anti-HBs Seroconversion Rate at Months 12
Anti-HBs Seroconversion Rate at Months 18 | Months 18
  Anti-HBs Seroconversion Rate at Months 18
Anti-HBs Seroconversion Rate at Months 24 | Months 24
  Anti-HBs Seroconversion Rate at Months 24
Anti-HBs Seroconversion Rate at Months 30 | Months 30
  Anti-HBs Seroconversion Rate at Months 30

SECONDARY OUTCOMES:
Anti-HBs Concentration at Months 1 | Months 1
  Anti-HBs Concentration at Months 1
Anti-HBs Concentration at Months 3 | Months 3
  Anti-HBs Concentration at Months 3
Anti-HBs Concentration at Months 7 | Months 7
  Anti-HBs Concentration at Months 7
Anti-HBs Concentration at Months 12 | Months 12
  Anti-HBs Concentration at Months 12
Anti-HBs Concentration at Months 18 | Months 18
  Anti-HBs Concentration at Months 18
Anti-HBs Concentration at Months 24 | Months 24
  Anti-HBs Concentration at Months 24
Anti-HBs Concentration at Months 30 | Months 30
  Anti-HBs Concentration at Months 30

OTHER OUTCOMES:
Occurrence of Adverse Events After Vaccination | Within 7 days after the vaccination
  Occurrence of Adverse Events After Vaccination
Occurrence of Adverse Events After Vaccination | Within 28 days after vaccination
  Occurrence of Adverse Events After Vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Suping Wang, PhD, Principal Investigator — Shanxi Medical University

IPD SHARING:
Plan to Share IPD: No